CLINICAL TRIAL: NCT00062569
Title: Reminiscence During Bathing Persons With Alzheimer's Disease at Home
Brief Title: Bathing Persons With Alzheimer's Disease aT Home (The BATH Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Ellen K. Mahoney, Boston College
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IA0044; R01NR007893-01A1 (NIH)
Record Dates: First submitted 2003-06-09; First posted 2003-06-12 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease; Resistiveness to baths; Caregiver stress; Bathing support intervention; Reminiscence; Agitated behavior; Resistiveness to care
MeSH Terms: conditions — Alzheimer Disease; Caregiver Burden; Psychomotor Agitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Bathing Support Intervention (BSI)
- 2 (Experimental)
  Interventions: Behavioral: Caregiver reminiscence with coaching

INTERVENTIONS:
Behavioral: Bathing Support Intervention (BSI) — Bathing Support Intervention - Review of caregiver current practices and perceptions and care recipient behavioral symptoms associated with bathing with pattern analysis based on observation; skill building for bathing and communication techniques; coaching for implementation
  Arms: 1
Behavioral: Caregiver reminiscence with coaching — BSI plus Reminiscence - BSI as above plus caregiver interview to ascertain pleasant long-term memories (e.g. stories, pictures, music) developed into a "crib sheet" for caregiver use conversationally prior to and during the bath
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of a 3-week reminiscence intervention applied during bathing persons with Alzheimer's disease (AD) in decreasing resistiveness to care (RTC), relieving patient discomfort, and improving spouse caregiver appraisals of burden, capabilities and confidence while bathing the patient. Reminiscence provides opportunities for the patient to feel good and recall pleasant memories, easily done by caregivers in a home setting. Home visits and telephone calls from trained nurses provide coaching and practice for caregivers for the preliminary phase of this study. Each couple will be enrolled in the study for approximately 9 weeks. The study will recruit 100 patient/spouse caregiver couples randomly divided into one of two groups: reminiscence with coaching, or bathing support (control). Bathing support will be provided to participants in both conditions including: individualized assessment; education regarding bathing techniques for people with dementia; and individualized problem solving. In addition to the bathing support intervention, participants in the experimental group will receive a pleasant memories interview and reminiscence script with coaching for implementation. Caregivers will keep a journal of their experiences in bathing the care recipient.

DETAILED DESCRIPTION:
Bath time is often distressing to persons with Alzheimer's disease (AD), leading to behavioral symptoms of resistiveness to care. Encountering these behaviors is distressing for caregivers, as well. Most studies of intervention for behavioral symptoms of AD have been done in nursing homes, but most care takes place in the home. The overall goal of this research is to improve the at-home bathing experience of both patients with AD and their spouse caregivers. This study builds on preliminary studies that: 1) developed observational measures of patient behaviors, and 2) developed and pilot tested the reminiscence during bathing intervention.

This randomized clinical trial will evaluate the effectiveness of a 3-week reminiscence intervention, applied during bathing persons with AD, in decreasing resistiveness to care (RTC), relieving patient discomfort, and improving spouse caregiver appraisals of burden, self-efficacy with bathing, and satisfaction. Reminiscence provides an intervention that draws on preserved individuality and memories, easily implemented by caregivers in a home setting. Home visits and telephone calls provide coaching and practice for caregivers in implementation. The sample includes 100 patient/spouse caregiver couples, randomized into one of two groups: reminiscence with coaching or bathing support (control).

Bathing support will be provided to participants in both conditions including: individualized assessment; education regarding bathing techniques for people with dementia; and individualized problem solving. In addition to the bathing support intervention, participants in the experimental group will receive a pleasant memories interview and reminiscence script with coaching for implementation. Using repeated measures design, observations will be made at baseline, post-intervention (5 weeks), and follow-up (8 weeks).

In the coaching/practicing/support phase of the study, caregivers will receive 1-hour home visits by a Nurse Interventionist (NI) for two weeks with caregiver practice and telephone support in between the in-home coaching/support visits. During the home visits, the NI will: (a) review the written reminiscence script and "crib sheet" with the spouse and role-model its use, (b) discuss instructions for delivering the reminiscence intervention to the patient immediately prior to and during the bath/shower, (c) teach the spouse to record patient behavior and intervention intensity using visual analog scales, and (d) review general approaches to bathing including a calm, unhurried approach, smiling, eye contact, brief description of what to expect, simple directions with time for the patient to respond, encourage patient participation, try not to respond to negative behaviors, praise for positive behaviors. Spouse caregivers will be encouraged to practice using the reminiscence intervention with every bath/shower for a 2-week period and to record the frequency of program implementation throughout the week on the data sheets.

ELIGIBILITY:
Inclusion:

* Have a diagnosis of probable Alzheimer's disease or a related disorder according to standard criteria.
* Have functional dependence in bathing;
* Demonstrate resistiveness to care during bathing;
* Live in the community in a home setting (house, apartment, condominium);
* Have a primary caregiver spouse or partner who lives with the care recipient and agrees to be in the study; and
* Have no anticipated admission for long term care within 3 months.
* Must be married couples or life partners living with Alzheimer's disease or related disorder living within a 15-mile radius of Boston College.
* Spouse or caregiver partner is the primary caregiver, including assistance with bathing.
* Women and minorities are encouraged to participate.

Exclusion:

* Severe concomitant medical conditions of patient or spouse.
* Not fluent in English.
* Couple resides in an institutional setting.
* Couple anticipates a significant change of living situation within three months.
* Couple does not meet the above inclusion criteria.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2002-09; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Care Recipient: Resistiveness to care; discomfort | Baseline, post 3-week intervention, and 3-week follow-up.
Caregiver: Self-efficacy; interactive behaviors | Baseline, post 3-week intervention, and 3-week follow-up.

SECONDARY OUTCOMES:
Caregiver burden & satisfaction | Baseline, post 3-week intervention, and 3-week follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen K. Mahoney, DNS, RN, Principal Investigator — Boston College, William F. Connell School of Nursing
Locations (1):
- Boston College, William F. Connell School of Nursing, Chestnut Hill, Massachusetts, United States

REFERENCES:
- [Background] Mahoney EK, Hurley AC, Volicer L, Bell M, Gianotis P, Hartshorn M, Lane P, Lesperance R, MacDonald S, Novakoff L, Rheaume Y, Timms R, Warden V. Development and testing of the Resistiveness to Care Scale. Res Nurs Health. 1999 Feb;22(1):27-38. doi: 10.1002/(sici)1098-240x(199902)22:13.0.co;2-t. PMID 9928961
- [Background] Moss SE, Polignano E, White CL, Minichiello MD, Sunderland T. Reminiscence group activities and discourse interaction in Alzheimer's disease. J Gerontol Nurs. 2002 Aug;28(8):36-44. doi: 10.3928/0098-9134-20020801-09. PMID 12219552
- [Background] Mahoney E, Volicer L, Hurley A. (2000). Managing Challenging Behaviors in Persons with Dementia. Baltimore, MD: Health Professions Press.